CLINICAL TRIAL: NCT00803231
Title: Follow-up Data of Patients Treated With XIGRIS® DROTRECOGIN ALFA (ACTIVATED) in France
Brief Title: Follow-up Data of Patients Treated With XIGRIS® in France
Status: Completed | Type: Observational
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Other Study IDs: 12401; F1K-FR-B009 (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-02

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Retrospective cohort: Patient treated with Xigris between January 2006 and November 2008.
- Prospective cohort: Patient treated with Xigris between November 2008 and November 2009.

SUMMARY:
The transparency commission wishes that the laboratory Lilly France sets up a follow-up study describing the conditions of use of Xigris® in France.

The purpose of this study is to describe the characteristics of the treated patients, the conditions of drug use, in particular the conditions of treatment initiation and the clinical development of the patients during normal clinical practice, in particular rate and cause of mortality within one month.

DETAILED DESCRIPTION:
The objectives of the study as defined by the specific requirements of Transparency Commission are as follows:

* To describe the characteristics of the patients treated with Xigris®

  * socio-demographic characteristics,
  * clinical profile
* To determine the conditions of use of Xigris®

  * To describe previous treatments,
  * To observe delay before Xigris® initiation,
  * To describe dose, duration of treatment,
  * To study the concomitant treatments and the associated treatments
* To describe the clinical evolution of the patients

  * To observe mortality after 1 month
  * To describe reasons of death

ELIGIBILITY:
Patients are eligible to be included in the study if they meet the following criteria

* Patients treated with Xigris® during the study period in intensive care units in France
* Patients with a minimum age of 18 years
* Patients who are presenting in the normal course of care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients treated with Xigris® between January 1st, 2006 and August 31st 2008 in intensive care units in France will be enrolled retrospectively, whereas all adult patients treated with Xigris® between September 1st, 2008 and September 1st, 2009 will be enrolled prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 1004 (Actual)
Dates: Start 2008-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Mortality | 28 and 31 days

SECONDARY OUTCOMES:
Severe bleeding events | 28 and 31 days
Length of hospital stay | 28 and 31 days

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon- fri 9AM-5PM eastern time (UTC/GMT- 5 hours,EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this study, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suresnes, France